CLINICAL TRIAL: NCT01058031
Title: Neural Correlates of PTSD Prevention With MBSR in Iraqi Veterans
Brief Title: Neural Correlates of PTSD Prevention With Mindfulness Based Stress Reduction (MBSR) in Iraqi Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bremner Merit 007
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Stress Disorders, Posttraumatic; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): MBSR
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Mindfulness Based Stress Reduction

SUMMARY:
The purpose of this study is to compare Mindfulness Based Stress Reduction to a supportive therapy control group.

ELIGIBILITY:
Inclusion Criteria:

* PTSD related to OEF/OIF service

Exclusion Criteria:

* History of brain injury

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
PTSD symptom level measured with the CAPS | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Doug Bremner, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States